CLINICAL TRIAL: NCT01707017
Title: The Effects of Low- and High-intensity Resistance Exercise on Force-velocity Characteristics in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: S53709
Record Dates: First submitted 2012-10-02; First posted 2012-10-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2011-11

CONDITIONS: Effects of Strength Training in Older Adults
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- High-load strength training (Active Comparator)
  Interventions: Other: Strength training
- Low-load strength training (Active Comparator)
  Interventions: Other: Strength training
- Low-load + moderate-load strength training (Active Comparator)
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training

SUMMARY:
The purpose of this study is to compare the impact of high- and low-intensity resistance exercise on force-velocity characteristics, muscle mass and inflammatory processes in older adults. As all training protocols are designed to end with maximal effort, effects are expected to be similar between groups.

ELIGIBILITY:
Inclusion Criteria:

* age 60 to 80 years

Exclusion Criteria:

* Knee or hip prothesis
* Systematic training
* Cardiovascular disease
* Acute lower back pain
* Dementia

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in force-velocity characteristics of knee extensors | Baseline, 12weeks, 6 months

OTHER OUTCOMES:
Change in muscle volume | Baseline, 12weeks, 6 months
Change in maximal strength (one repetition maximum) | Baseline, 4weeks, 8weeks, 12weeks, 6 months
  Strength is measured as the maximum weight on the training equipment that can be lifted only one time (= one repetition maximum).
Change in motivation | Baseline, every week for 12 weeks, 6 months
Change in physical activity | Baseline, 12weeks, 6 months
Change in inflammatory markers in blood | Baseline, 12weeks, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Van Roie E, Walker S, Van Driessche S, Baggen R, Coudyzer W, Bautmans I, Delecluse C. Training load does not affect detraining's effect on muscle volume, muscle strength and functional capacity among older adults. Exp Gerontol. 2017 Nov;98:30-37. doi: 10.1016/j.exger.2017.07.017. Epub 2017 Aug 1. PMID 28778747
- [Derived] Nuvagah Forti L, Van Roie E, Njemini R, Coudyzer W, Beyer I, Delecluse C, Bautmans I. High Versus Low Load Resistance Training: The Effect of 24 Weeks Detraining on Serum Brain Derived-Neurotrophic Factor (BDNF) in Older Adults. J Frailty Aging. 2017;6(1):53-58. doi: 10.14283/jfa.2017.2. PMID 28244559